CLINICAL TRIAL: NCT03030924
Title: Physiologic Parameters for Monitoring Adolescent Suicidality
Brief Title: Wearable Suicidal Early Warning System for Adolescents
Status: Active, not recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dr. David Sheridan, Assistant Professor of Emergency Medicine/Pediatrics, Oregon Health and Science University
Other Study IDs: STUDY00016409; 5K12HL133115 (NIH)
Record Dates: First submitted 2017-01-21; First posted 2017-01-25 (Estimated); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Suicide; Adolescent Behavior
Keywords: suicide
MeSH Terms: conditions — Suicide; Adolescent Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Solace — Noninvasive physiologic monitor

SUMMARY:
This study is prospectively enrolling a cohort of adolescent patients who present to the Emergency Department and an inpatient psychiatric adolescent unit with acute suicidality.

DETAILED DESCRIPTION:
This study is prospectively enrolling a cohort of adolescent patients who present to the Emergency Department with acute suicidality or are admitted to an inpatient psychiatric adolescent unit. The plan is to monitor basic physiologic parameters to assess for trends associated with suicidality noninvasively in an objective manner beyond subjective questionnaires currently available. Upon discharge they will be sent home with a noninvasive monitor to track physiologic parameters.

ELIGIBILITY:
Inclusion Criteria:

* acute suicidality
* consenting individual present in the emergency department

Exclusion Criteria:

* medical admission for an ingestion or other reason

Ages: 13 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents presenting with acute suicidal thoughts or attempts in the pediatric emergency department (13-19 years of age).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-09-18 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | 1 week

SECONDARY OUTCOMES:
Gender | At enrollment
Age | at enrollment
  in Years
Columbia Suicide Severity Score | 1 week
  Numerical based on severity
PHQ-9 Depression Scale | 1 week
  Numerical based on severity
Motion | 1 week
  As detected by an accelerometer in Hz

OTHER OUTCOMES:
past Medical History | At enrollment
Medications | At enrollment and daily for one week after discharge
  Daily medications

CONTACTS AND LOCATIONS:
Overall Officials: David Sheridan, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheridan DC, Lin A. Emergency Department Adolescent Suicidality: A Pilot Study to Determine How Common Actual Attempts Are. Pediatr Emerg Care. 2022 Feb 1;38(2):e458-e461. doi: 10.1097/PEC.0000000000002629. PMID 35100750
- [Derived] Sheridan DC, Dehart R, Lin A, Sabbaj M, Baker SD. Heart Rate Variability Analysis: How Much Artifact Can We Remove? Psychiatry Investig. 2020 Sep;17(9):960-965. doi: 10.30773/pi.2020.0168. Epub 2020 Sep 18. PMID 33017533